CLINICAL TRIAL: NCT06283004
Title: The Effect of Aerobic Exercise Training in Different Slope Types on Exercise Capacity, Respiratory Functions, Muscle Strength, and Functional Status in COPD Patients
Brief Title: Investigation of Walking Training With Different Slope Types in COPD Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Collaborators: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Meryem BEKTAŞ KARAKUŞ, Research Assistant, Principal Investigator, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1/30
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Level walking (Active Comparator): It will walk at a 0-degree slope (0) throughout the research.
  Interventions: Other: Level walking training
- Downhill walking (Experimental): It will walk at a 10-degree downhill slope (-10) throughout the research.
  Interventions: Other: Downhill walking training
- Uphill walking (Experimental): It will walk at a 10-degree uphill slope (+10) throughout the research.
  Interventions: Other: Uphill walking training

INTERVENTIONS:
Other: Downhill walking training — For 8 weeks, downhill walking training will be done 2 times a week at a slope of -10 degrees.
  Arms: Downhill walking
Other: Level walking training — For 8 weeks, level walking training will be done 2 times a week at a slope of 0 degrees.
  Arms: Level walking
Other: Uphill walking training — For 8 weeks, uphill walking training will be done 2 times a week at a slope of +10 degrees.
  Arms: Uphill walking

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a disease that continues to generate a great deal of research and this research must continue, both because it is not completely curable and because of the large patient population. The importance and benefits of exercise training in COPD patients are clear. One of the most preferred types of exercise training is the so-called aerobic exercise training, which typically takes the form of walking. A typical walking training does not use a slope or may include an uphill slope. However, recently there have been publications about downhill walking and its benefits in COPD. Walking on a level, uphill, and downhill slope may have the potential to result in different gains by using different muscle groups more. Therefore, this study aimed to compare the effects of walking training on exercise capacity, respiratory functions, muscle strength, and functional status in COPD patients with three different slope types: level, uphill, and downhill.

DETAILED DESCRIPTION:
The convenience sampling method will be used as the sampling method in the research.

In this study, sample size was calculated by a priori power analysis using G*Power 3.1.9.4 software. In the analysis for analysis of variance (ANOVA: repeated measures, between factors) with two factors and repeated measures; effect size f = 0.62 (based on data obtained from previous study, Borghi-Silva et al, 2009), significance level α = 0.05, statistical power (1 - β) = 0.80, number of groups 3, number of measures 2 and correlation coefficient between measures r = 0.5. According to the calculation, it was predicted that the study would reach sufficient statistical power with a total of 24 participants, 8 participants in each group.

There will be three groups in the study: downhill walking, uphill walking, and level walking. The downhill walking and uphill walking groups will be included as the study group and the level walking group will be included as the control group. Participants will be distributed equally to the three groups. Patients will be assigned to these groups by block randomization method using https://www.randomizer.org/ website.

All three groups will be administered a 6-minute walking test at baseline, and participants will be subjected to a common 8-week, twice-weekly treadmill walking training program in which the speed is determined and increased according to the average speed they walk in this test, and in addition to this, the duration is also increased. One session of the training program will consist of warming up, loading, and cooling down on the treadmill.

During the training, the slope of the treadmill will be adjusted to +10 degrees for uphill walking, -10 degrees for downhill walking, and 0 degrees for level walking and will be kept constant for 8 weeks. A special wooden wedge apparatus will be made under the normal treadmill to give -10 downhill slope.

Primary outcome measurements will be made at baseline and at the end of week 8.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with COPD (A, B, E groups according to GOLD assessment)
* Ambulate on your own
* Not having any contraindications for exercise
* To be mentally appropriate (score 24 points and above in the mini mental test)

Exclusion Criteria:

* Being in GOLD 4 stage in spirometric evaluation
* Presence of hypoxemia
* Participation in another pulmonary rehabilitation program within the last 6 months
* Having an exacerbation in the last 1 month
* Being diagnosed with additional respiratory disease (asthma, bronchiectasis, etc.)
* Having had pulmonary surgery
* Having an orthopedic, neurological or cardiac disease that affects exercise
* Having uncontrolled hypertension or diabetes
* Presence of malignancy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2025-04-09 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
6 Minutes Walking Distance (6MWD) | Up to 8 weeks.
  6 MWD means the distance traveled in 6 MWT. Its unit is meters.
Spirometric measurements (Forced vital capacity) | Up to 8 weeks.
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. Forced vital capacity (FVC): the maximum amount of air that can be forcibly exhaled from the lungs after fully inhaling. It can be recorded in percentages or liters.
Spirometric measurements (First second forced expiratory volume) | Up to 8 weeks.
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. First-second forced expiratory volume (FEV1): the amount of air that can be exhaled with force in 1 second. It can be recorded in percentages or liters.
Spirometric measurements (FEV1/FVC ratio) | Up to 8 weeks.
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. It is calculated by dividing FEV1 by FVC. It is expressed as a percentage.
Spirometric measurements (Peak Expiratory Flow) | Up to 8 weeks.
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. Peak expiratory flow (PEF) is the maximum flow achieved during a forced expiration starting from the level of maximal lung inflation. It can be recorded in percentages or liters.
Spirometric measurements (Maximum Intermediate Expiratory Flow) | Up to 8 weeks.
  It is used to evaluate respiratory functions. It is evaluated with a spirometer. Maximum Intermediate Expiratory Flow (FEF25-75) is the flow (or speed) of air coming out of the lung during the middle portion of a forced expiration. It can be recorded in percentages or liters.
Muscle strength measurements (skeletal muscles) | Up to 8 weeks.
  Hip extension, knee extension, and ankle extension muscle strength will be measured with a handheld dynamometer. The results are recorded in Newtons.
Muscle strength measurements (respiratory muscles) | Up to 8 weeks.
  The strength of the respiratory muscles will be assessed and recorded as maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) with a device that allows the measurement of intraoral pressures, which is an indirect indicator of the strength of these muscles. In this device, measurements are based on recording the highest average pressure sustained for one second during inspiration and expiration against a closed valve. Measurements are recorded in cmH2O.
30-second sit and stand test | Up to 8 weeks.
  The result is the total number of stands within 30 seconds.
Functional performance inventory | Up to 8 weeks.
  It is a valid and reliable measurement tool used to assess functional performance in COPD patients. It consists of 6 sub-dimensions (body care, household maintenance, physical exercise, recreation, spiritual activities, social activities) and a total of 65 items. The questions are answered by choosing from the following options: "I can do the activity easily without any difficulty (3 points), I can do it with some difficulty (2 points), I can do it with much difficulty (1 point), I can no longer do this activity due to my health reasons (0 points), I do not prefer it (0 points)" and are scored according to the specified scores. Each sub-dimension and total performance is calculated as an average. The lowest score is 0 and the highest score is 3. Higher score means better functional performance. Turkish validation study of the questionnaire in COPD patients was conducted.

SECONDARY OUTCOMES:
Dyspnea | Up to 8 weeks.
  It will be reported by the participant using the modified borg scale (between 0-10 points). On this scale, 0 is the lowest score and means absent, while 10 is the highest score and indicates that the condition is most severe.
Fatigue | Up to 8 weeks.
  It will be reported by the participant using the modified borg scale (between 0-10 points).On this scale, 0 is the lowest score and means absent, while 10 is the highest score and indicates that the condition is most severe.
Level of exertion | Up to 8 weeks.
  It will be reported by the participant using the modified borg scale (between 0-10 points). On this scale, 0 is the lowest score and means absent, while 10 is the highest score and indicates that the condition is most severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Department of Physiotherapy and Rehabilitation, Istanbul, Eyüp Sultan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borghi-Silva A, Arena R, Castello V, Simoes RP, Martins LE, Catai AM, Costa D. Aerobic exercise training improves autonomic nervous control in patients with COPD. Respir Med. 2009 Oct;103(10):1503-10. doi: 10.1016/j.rmed.2009.04.015. Epub 2009 May 22. PMID 19464865
- [Background] Vallera DA, Blazar BR. Depressed leukocyte reconstitution and engraftment in murine recipients of T cell-depleted histoincompatible marrow pretreated with interleukin 3. Transplantation. 1988 Oct;46(4):616-20. doi: 10.1097/00007890-198810000-00039. No abstract available. PMID 3262943
- [Background] Alexander N, Strutzenberger G, Ameshofer LM, Schwameder H. Lower limb joint work and joint work contribution during downhill and uphill walking at different inclinations. J Biomech. 2017 Aug 16;61:75-80. doi: 10.1016/j.jbiomech.2017.07.001. Epub 2017 Jul 11. PMID 28734544
- [Background] Nordback I, Lauslahti K. Clinicopathologic and histochemical study of ovarian clear cell carcinoma. Int J Gynaecol Obstet. 1980 Sep-Oct;18(2):85-9. doi: 10.1002/j.1879-3479.1980.tb00251.x. PMID 6108258
- [Background] Camillo CA, Burtin C, Hornikx M, Demeyer H, De Bent K, van Remoortel H, Osadnik CR, Janssens W, Troosters T. Physiological responses during downhill walking: A new exercise modality for subjects with chronic obstructive pulmonary disease? Chron Respir Dis. 2015 May;12(2):155-64. doi: 10.1177/1479972315575717. Epub 2015 Mar 10. PMID 25758676
- [Background] Brooks RG. Postgraduate training in child psychiatry: the content of the curriculum. Am J Psychiatry. 1973 Apr;130(4):491-3. doi: 10.1176/ajp.130.4.491. No abstract available. PMID 4691311
- [Background] Camillo CA, Osadnik CR, Burtin C, Everaerts S, Hornikx M, Demeyer H, Loeckx M, Rodrigues FM, Maes K, Gayan-Ramirez G, Janssens W, Troosters T. Effects of downhill walking in pulmonary rehabilitation for patients with COPD: a randomised controlled trial. Eur Respir J. 2020 Sep 17;56(3):2000639. doi: 10.1183/13993003.00639-2020. Print 2020 Sep. PMID 32444407
- [Background] Leidy NK. Psychometric properties of the functional performance inventory in patients with chronic obstructive pulmonary disease. Nurs Res. 1999 Jan-Feb;48(1):20-8. doi: 10.1097/00006199-199901000-00004. PMID 10029398